CLINICAL TRIAL: NCT01687894
Title: Clinical Trials of Vasopressin for Prevention of Hypotension During Shoulder Surgery in Beach Chair Position Under General Anesthesia
Brief Title: Vasopressin to Prevent Hypotension During Beach Chair Surgery
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Chonnam National University (Other)
Responsible Party: Principal Investigator, Kyung Yeon Yoo, Professor, Chonnam National University Hospital
Other Study IDs: CNUH-2012-074
Record Dates: First submitted 2012-09-08; First posted 2012-09-19 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2012-09

CONDITIONS: Rotator Cuff Tear Arthropathy
Keywords: cerebral oxygen saturation; beach chair position; hemodynamic; jugular venous oximetry
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy | interventions — Vasopressins; Arginine Vasopressin; Sodium Chloride; Propofol; Anesthetics, Intravenous; Sevoflurane; Anesthetics, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Vasopressins & propofol: Administer vasopressin 0.05 or 0.07 IU/kg before sitting position during propofol anesthesia.
  Interventions: Drug: Vasopressins; Drug: propofol
- Placebo & propofol: Administer saline 10 ml (placebo) 2 min before beach chair position during propofol anesthesia
  Interventions: Drug: Placebo; Drug: propofol
- Vasopressins & sevoflurane: Administer vasopressin 0.05 or 0.07 IU/kg 2 min before beach chair position during sevoflurane anesthesia
  Interventions: Drug: Vasopressins; Drug: sevoflurane
- Placebo & sevoflurane: Placebo (saline 10 ml) for vasopressin is administered 2 min before beach chair position during sevoflurane anesthesia
  Interventions: Drug: Placebo; Drug: sevoflurane

INTERVENTIONS:
Drug: Vasopressins — Vasopressins propofol vasopressins sevoflurane
  Other Names: Arginine vasopressin
  Groups: Vasopressins & propofol; Vasopressins & sevoflurane
Drug: Placebo — Placebo propofol & placebo sevoflurane
  Other Names: saline 10 ml as placebo
  Groups: Placebo & propofol; Placebo & sevoflurane
Drug: propofol — vasopressin propofol & placebo propofol
  Other Names: Intravenous anesthetic
  Groups: Placebo & propofol; Vasopressins & propofol
Drug: sevoflurane — vasopressins sevoflurane placebo sevoflurane
  Other Names: general anesthetic
  Groups: Placebo & sevoflurane; Vasopressins & sevoflurane

SUMMARY:
Patients undergoing surgery in beach chair position (BCP) are at risk for cerebral ischaemia. The impacts of arginine vasopressin (AVP) on haemodynamics and cerebral oxygenation are evaluated during surgery in BCP.

DETAILED DESCRIPTION:
Patients undergoing shoulder surgery in BCP under general anaesthesia are randomly allocated to receive i.v. normal saline (control group) or AVP 0.05 or 0.07 U kg-1 (AVP group, n = 15 each) 2 min before moving into BCP. Mean arterial pressure (MAP), heart rate (HR), jugular venous bulb oxygen saturation (SjvO2) and regional cerebral tissue oxygen saturation (SctO2) are measured before (pre-sitting in supine position) and after patients assumed BCP.

ELIGIBILITY:
Inclusion Criteria: elective arthroscopic shoulder surgery under general anesthesia in beach chair position

Exclusion Criteria: preexisting cerebrovascular diseases, history of orthostatic hypotension, age less than 18 yr, and the American Society of Anesthesiologists physical status IV or V

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing shoulder surgery in the beach chair position under the general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The magnitude of decrease of mean arterial pressure | Baseline (before positioning) and lowest value within 10 min into beach chair position
  Continuously measure mean arterial blood pressure before and after position change. Calculate the magnitude of maximum decrease of mean arterial pressure from baseline

SECONDARY OUTCOMES:
Jugular venous oxygen desaturation | Up to 30 min after the positioning
  Jugular venous oxygen saturation is continuously measured whether its saturation is decreased below 50% or/and 40% for longer than 5 min.

OTHER OUTCOMES:
Cerebral oxygen desaturation | Up to 30 min after the position change
  Continuously observe near-infrared spectroscopy measured cerebral oxygenation before and after beach chair position whether oxygen saturation decrease more than 20% from pre-sitting values

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Y Yoo, M.D.,Ph.D, Principal Investigator — Department of Anesthesiology and Pain Medicine, Chonnam National University Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Gwangju, South Korea

REFERENCES:
- [Derived] Jang EA, Song JA, Shin JY, Yoon JJ, Yoo KY, Jeong S. Background anaesthetic agents do not influence the impact of arginine vasopressin on haemodynamic states and cerebral oxygenation during shoulder surgery in the beach chair position: a prospective, single-blind study. BMC Anesthesiol. 2017 May 30;17(1):73. doi: 10.1186/s12871-017-0364-9. PMID 28558702